CLINICAL TRIAL: NCT04448119
Title: Control of COVID-19 Outbreaks in Long Term Care (CONTROL-COVID)
Brief Title: Control of COVID-19 Outbreaks in Long Term Care
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: Appili Therapeutics Inc. (Industry)
Collaborators: MOUNT SINAI HOSPITAL (Other); Applied Health Research Centre (Other); Sunnybrook Health Sciences Centre (Other); University Health Network, Toronto (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CONTROL-COVID-Favipiravir-1
Record Dates: First submitted 2020-06-24; First posted 2020-06-25 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: COVID-19; Long-Term Care Home; Favipiravir; Chemoprophylaxis; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — favipiravir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemoprophylaxis (Experimental): Participants of LTCH units allocated to the chemoprophylaxis arm receive favipiravir for 25 days. Residents in the LTCH unit diagnosed with COVID- 19 at enrollment will be offered treatment with favipiravir for 14 days.
  Interventions: Drug: Favipiravir
- Placebo (Placebo Comparator): Participants of LTCH units allocated to the control arm receive placebo for 25 days. Residents in the LTCH unit diagnosed with COVID-19 at enrollment will be offered treatment with placebo for 14 days.
  Interventions: Drug: Favipiravir Placebo

INTERVENTIONS:
Drug: Favipiravir — Favipiravir is the experimental drug. The dosage for favipiravir to be used in this study for prophylaxis is 1600 mg (8 x 200 mg tablets) orally twice daily on day 1 followed by 800 mg (4 x 200 mg tablets) orally twice daily on days 2-25. The dose of favipiravir for treatment is 2000 mg orally twice daily on day 1, the 1000 mg orally twice daily for 13 additional days.
  Other Names: Avigan
  Arms: Chemoprophylaxis
Drug: Favipiravir Placebo — Favipiravir Placebo is the placebo drug. For chemoprophylaxis, the dosage of favipiravir placebo is 8 tablets orally twice daily on day 1, followed by 4 tablets twice daily from days 2-25. The dosage of favipiravir placebo for treatment is 10 tablets orally twice daily on day 1, followed by tablets twice daily from days 2-14.
  Arms: Placebo

SUMMARY:
To address the need to intervene to prevent the spread of COVID-19 in long-term care homes, we propose a randomized clinical trial of chemoprophylaxis in long-term care homes experiencing COVID-19 outbreaks. LTCH units experiencing an outbreak of COVID-19 will be randomized to chemoprophylaxis with favipiravir or placebo in a 1:1 ratio.

Chemoprophylaxis in this setting refers to the use of favipiravir for pre-exposure prophylaxis, post-exposure prophylaxis, pre-emptive therapy, or treatment for established COVID-19. This design mimics the approach to influenza outbreaks, which has proven efficacy for outbreak control. The primary outcome will be control of the outbreak, defined as no new microbiologically confirmed case of COVID-19 for 24 consecutive days up to day 40.

DETAILED DESCRIPTION:
Early in the COVID-19 pandemic, it became apparent that the elderly are disproportionately bearing the burden of disease and mortality. Many outbreaks are occurring in long-term care homes (LTCHs), with strikingly high mortality rates: nearly two-thirds of all Canadian COVID- 19 deaths are in LTCH residents. This is unsurprising, as viral respiratory outbreaks in LTCHs are devastating: before the use of influenza vaccine, case fatality rates during influenza outbreaks were as high as 55%. Interventions are thus urgently needed to control LTCH outbreaks to mitigate harms to this vulnerable population and maximize acute care capacity.

Chemoprophylaxis is the cornerstone of management of LTCH influenza outbreaks and disease prophylaxis has been deemed a critical COVID-19 research priority by the World Health Organization. While definitive therapies do not yet exist, there is significant interest in repurposing existing anti-viral agents against COVID-19. Favipiravir, a broad spectrum antiviral agent, demonstrates activity against SARS-CoV-2 in vitro, and was associated with faster viral clearance, radiographic improvement, and clinical recovery in early trials. Favipiravir is an ideal candidates for chemoprophylaxis, as it is orally available and has a reasonable safety profile.

To address the need to intervene to prevent the spread of COVID-19 in LTCHs, we propose a cluster-randomized placebo-controlled trial of chemoprophylaxis in LTCHs experiencing COVID-19 outbreaks.

This study is a partially blinded, placebo-controlled cluster randomized trial of chemoprophylaxis to control outbreaks of COVID-19 in LCTHs for the elderly. The unit of analysis is a ward/unit. An outbreak is defined as ≥ 2 symptomatic microbiologically-confirmedCOVID-19 cases within 7 days on the LTCH unit. This design is selected to mimic the current approach to outbreaks of other respiratory viral infections, both because this approach has proven effective for these other viruses, and because it is standard practice and therefore feasible to implement.

Eligible LTCHs will be asked to report outbreaks to the study in addition to the legally-required reporting to their local public health unit; public health units will also be asked to discuss the study with LTCHs reporting outbreaks. In addition, study staff will contact the infection control practitioner in each of the screened LTCHs twice weekly, to ensure the prompt identification of outbreak units.

Residents and staff will be assessed for contraindications to enrollment and informed consent will be obtained for residents and staff to receive the allocated intervention, and to be followed up individually for clinical outcomes, adherence and safety during the outbreak.

LTCH units experiencing an outbreak of COVID-19 will be randomized to either favipiravir or placebo in a 1:1 ratio. Favipiravir or placebo will be offered to all residents and staff who will be working on the unit during the chemoprophylaxis period, according to the allocation. Study drug will continue for a duration of 25 days. The dosage for favipiravir to be used in this study for chemoprophylaxis is 1600 mg (8 x 200 mg tablets) orally twice daily on day 1 followed by 800 mg (4 x 200 mg tablets) orally twice daily on day 2-25. Residents in the LTCH unit diagnosed with COVID-19 at enrollment will be offered treatment with favipiravir or placebo for 14 days, according to the LTCH unit allocation. The dose of favipiravir for treatment is 2000mmg orally twice daily on day 1, then 1000 mg orally twice daily for 13 additional days.

Surveillance for infection will occur as usual for resident illness within each LTCH; staff will be asked to report symptoms and will be screened for symptoms each time they enter the building. Consenting residents and staff will be screened at day 0, day 14 and day 40 to identify asymptomatic infections and to assess duration of viral shedding. The primary outcome will be control of the outbreak, defined as no new microbiologically confirmed case of COVID-19 for 24 consecutive days up to day 40.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for LTCHs:

  1. LTCH in Ontario with >80% of residents being adults ≥65 years of age.
  2. Residents are or can be routinely assessed at least daily by staff.
  3. LTCH has not previously had a unit enrolled in this study.
  4. Outbreak of COVID-19 declared on at least one nursing unit, requiring all of the following:

     1. ≥2 to ≤4 residents who develop PCR-confirmed symptomatic COVID-19 infection on the same unit within ≤ 7 days at the time when the outbreak is identified as eligible.
     2. ≤21 days from symptom onset in the index case at the time when the outbreak is identified as eligible.
     3. Cumulative attack rate in residents on the affected unit since the beginning of the pandemic ≤25% at the time when the outbreak is identified as eligible.
     4. ≤20% of residents with microbiologically confirmed COVID-19 or line-listed as a presumptive case in a COVID-19 outbreak and not tested for COVID-19 in prior outbreaks within the last six months.
     5. Nursing unit with ≥16 and ≤32 residents.
     6. Nursing home agrees to work with study coordination to minimize the number of persons who provide care on the unit.
  5. Mechanism exists for delivery of medication and recording of administered medication for all residents.
  6. ≥80% of residents on outbreak unit are eligible and they or their substitute decision makers consent to participate in the study.
  7. Written informed consent of Medical Director, Administrator and a delegate of the Residents' Council of the LTCH for LTCH to be included in the cluster trial.
* Inclusion criteria for LTCH residents:

  1. Informed consent from resident or substitute decision maker (SDM)
* Inclusion criteria for LTCH staff:

  1. Expected to work at least two 8-hour shifts, or the equivalent time (16 hours on the unit) during the outbreak period.
  2. Informed consent.

Exclusion Criteria:

* Exclusion criteria for LTCHs:

  1. Inability to deliver medication to consenting residents within 96 hours of identification of the outbreak.
  2. Inability to define a physically separate unit with ≤32 residents.
  3. Any of facility management, medical advisory committee or resident council do not approve participation.
* Exclusion criteria for LTCH Residents and Staff:

  1. Pregnancy (females < 55 years of age require a negative urine pregnancy test at enrollment, and either menopause or two concurrent reliable methods of contraception need to be confirmed)
  2. History of abnormalities of uric acid metabolism, other than gout.
  3. History of hypersensitivity to remdesivir or favipiravir
  4. Previous diagnosis of hepatic cirrhosis
  5. Current use of the following medications, which cannot be discontinued for the duration of the study: pyrazinamide, hydralazine, more than 3000 mg of acetaminophen per day

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Control of Outbreak | Day 40
  Control of outbreak, defined as no new cases of COVID-19 in residents for 24 consecutive days up to day 40 after the start of prophylaxis

SECONDARY OUTCOMES:
Mortality (Residents) | Day 40, Day 60
  The proportion of residents of included LTCH units who die up to day 40, and up to day 60
COVID-19 Infection (Residents) | Day 40
  The proportion of residents of included LTCH units who were uninfected at baseline and develop new symptomatic microbiologically confirmed COVID-19 up to day 40
COVID-19 Infection (Staff) | Day 14, Day 40
  The proportion of exposed staff uninfected at baseline in whom SARS-CoV-2 infection is identified up to day 14 and up to day 40
Hospitalization (Residents) | Day 40
  The proportion of residents of included LTCH units hospitalized up to day 40
Medication Discontinuation (Residents) | Day 40
  The proportion of residents of included LTCH units who discontinue study medication due to adverse events
Medication Discontinuation (Staff) | Day 40
  The proportion of LTCH staff of included LTCH units who discontinue study medication due to adverse events
COVID-19 in new LTCH Units (a) | Day 40
  The occurrence of new microbiologically confirmed COVID-19 infections in residents in other units of the LTCH up to day 40 (dichotomous, at LTCH level)
COVID-19 in new LTCH Units (b) | Day 40
  The proportion of previously unaffected LTCH units of the remainder of the LTCH in which a case of COVID-19 is identified
COVID-19 in new LTCH Units (c) | Day 40
  The proportion of residents in the remainder of the LTCH who develop COVID-19 infections up to day 40

CONTACTS AND LOCATIONS:
Overall Officials: Allison J McGeer, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No